CLINICAL TRIAL: NCT05408637
Title: Transcranial Photobiomodulation for Executive Function in Bipolar Disorder (TPEB)
Brief Title: Transcranial Photobiomodulation for Executive Function in Bipolar Disorder
Acronym: TPEB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Paolo Cassano (Other)
Responsible Party: Sponsor-Investigator, Paolo Cassano, Director of Photobiomodulation, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2022p000289
Record Dates: First submitted 2022-05-17; First posted 2022-06-07 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Bipolar Disorder
Keywords: Bipolar; Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: All participants will receive five active tPBM treatments and one sham tPBM treatment.
Who Masked: Participant
Masking Description: During the first treatment visit within the MRI, participants will receive one active tPBM treatment and one sham tPBM treatment. Participants will be blinded as to the order in which they receive these treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Transcranial Phoobiomodulation (tPBM) — Transcranial light therapy penetrates the skin and brain using light energy; this makes transcranial light therapy noninvasive. Transcranial light therapy may activate under-stimulated brain regions.
  Other Names: Transcranial Light Therapy; Low Level Laser-Light Therapy

SUMMARY:
Transcranial light therapy, or transcranial photobiomodulation (tPBM), is a treatment that stimulates the brain by applying near-infrared light to the forehead. Transcranial light therapy has been found to promote brain metabolism, which may help improve executive function in people with bipolar disorder. The research team proposes a novel approach to treating bipolar disorder by using transcranial light therapy.

DETAILED DESCRIPTION:
This study involves a virtual screening visit, 7 in-office visits, and a virtual check-in call with a clinician. Participation will last approximately 3 weeks in total.

Participants will attend a baseline visit during which they will complete mood questionnaires and a gambling task. Participants will then receive five treatments of transcranial light therapy over one week. The first and last of these treatments will be administered while the participant is in an MRI scanner. At the first visit, participants will also receive a "sham" tPBM treatment, meaning that the device will simulate real treatment, but will not actually apply the near-infrared light. The check-in call will occur approximately 2-3 days after the final treatment visit. This will be a brief call with a study clinician to check-in on the participant's mental and physical health. The follow up visit will occur approximately one week after the final visit. Subjects will be asked to complete mood questionnaires and/or gambling tasks during the first and fifth treatment visits, as well as at the follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18 and 65
* Diagnosis of bipolar disorder
* Currently experiencing symptoms of impulsivity
* Vision normal or corrected to normal with contacts

Exclusion Criteria:

* Currently in depressive, manic, or mixed episode
* Currently psychotic
* Judged to be at serious and imminent suicidal risk
* Currently in alcohol or substance use disorder (meeting criteria in the past 3 months)
* Unstable medical conditions
* Inability to consent or to complete study procedures
* Failure to meet standard MRI safety requirements (e.g. claustrophobia, non-removable piercings, implanted medical devices, other non-removable metals)
* Changes in medications or use of augmentative devices and other interventions in the 2 weeks prior to the study
* Participation in other clinical research trials that may influence primary outcomes or adherence to the proposed study
* Current pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mass General Hospital Navy Yard Building 149, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at Massachusetts General Hospital between July 2022 and April 2024. Subjects were recruited through a variety of methods, including online advertisements and surveys, flyers, and referrals from providers and other research studies.
Pre-assignment Details: Subjects underwent screening procedures to determine eligibility. A majority of subjects were excluded for not meeting the impulsivity threshold. Other subjects were excluded due to current alcohol or substance use disorder or were lost to follow up.
Groups:
- Transcranial Light Therapy: Subjects who passed screening and completed all study procedures.
  All subjects received a sham light therapy treatment followed by an active light therapy treatment at the first MRI session. This was a single-blind procedure. All following transcranial photobiomodulation (tPBM) sessions (Treatment Days 2, 3, 4 and MRI session on Day 5) were active and open-label.
Period: Overall Study
Arm/Group | Transcranial Light Therapy
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Subjects: Subjects who passed screening and completed all study procedures.
Arm/Group | Subjects
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (4.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4
Barrat Impulsiveness Scale (BIS) [Mean (Standard Deviation); unit: units on a scale] — Measure of impulsivity. Higher scores indicate higher impulsivity (min 30, max 120, lower score=better outcome)
  units on a scale | 69.75 (8.77)

OUTCOME MEASURES:

1. Primary Outcome: Test the Effect of Transcranial Photobiomodulation (tPBM) on Cerebral Blood Flow (CBF)
Description: Compare blood-oxygenation-level-dependent (BOLD) signal during sham stimulation at Day 1 versus BOLD signal during active stimulation at Day 1. Increased BOLD signal is thought to reflect increased brain activity, and thus a positive outcome. In this specific case, higher BOLD signal during active as compared to sham treatment in the right dorsolateral prefrontal cortex (rDLPFC) is thought to reflect target engagement, that is the tPBM device which is placed on the right forehead is in fact irradiating and having an effect on brain function within the rDLPFC.
Time Frame: Day 1 of tPBM Treatment
Measure: Mean (Standard Deviation); unit: A.U.
Groups:
- Transcranial Light Therapy Subjects: Subjects who passed screening and completed all study procedures.
  All subjects received a sham light therapy treatment followed by an active light therapy treatment at the first MRI session. This was a single-blind procedure.
Arm/Group | Transcranial Light Therapy Subjects
Number analyzed (Participants) | 4
A.U.
  Sham Stimulation BOLD Signal | 6611.645 (794.5616)
  Active Stimulation BOLD Signal | 6666.398 (784.01)
Statistical Analysis 1: Comparison: Transcranial Light Therapy Subjects; Test type: Other — The small sample size did not allow for statistical tests. Therefore, we looked at overall patterns and calculated differences between stimulation (Active vs Sham); Mean Difference (Final Values) = 54.75 — Difference = Active - Sham
Statistical Analysis 2: Comparison: Transcranial Light Therapy Subjects; The small sample size did not allow for statistical tests. Therefore, we looked at percent difference between stimulation (Active vs Sham); Test type: Other; Percent Difference = 0.85 — Difference = Active - Sham
Statistical Analysis 3: Comparison: Transcranial Light Therapy Subjects; We evaluated the effect size of the difference between Active and Sham using Cohen's d; Test type: Other; Cohen's d = 0.07

2. Primary Outcome: Test Effect of tPBM on CBF
Description: Compare BOLD signal during active stimulation at Day 1 versus active stimulation at Day 5. Greater BOLD signal at Day 5 compared to Day 1 would indicate an increase in brain activity following active treatment, supporting tPBM target engagement.
Time Frame: Day 1 and Day 5
Measure: Mean (Standard Deviation); unit: A.U.
Groups:
- Transcranial Light Therapy Subjects: Subjects who passed screening and completed all study procedures.
  All subjects received active tPBM Days 1-5. The first treatment on Day 1 was single-blind, all others were open-label.
Arm/Group | Transcranial Light Therapy Subjects
Number analyzed (Participants) | 4
A.U.
  Day 1 Active BOLD Signal | 6666.398 (784.01)
  Day 5 Active BOLD Signal | 6891.237 (412.7808)
Statistical Analysis 1: Comparison: Transcranial Light Therapy Subjects; Test type: Other — The small sample size did not allow for statistical tests. Therefore, we looked at overall patterns and calculated differences between active stimulation timepoints (Day 1 vs Day 5); Mean Difference (Final Values) = 224.8392 — Difference = Day 5 Active - Day 1 Active
Statistical Analysis 2: Comparison: Transcranial Light Therapy Subjects; The small sample size did not allow for statistical tests. Therefore, we calculated percent difference between active stimulation timepoints (Day 1 vs Day 5); Test type: Other; Percent Difference = 4.35 — Difference = Day 5 Active - Day 1 Active
Statistical Analysis 3: Comparison: Transcranial Light Therapy Subjects; We evaluated the effect size of the difference between active stimulation timepoints (Day 1 vs Day 5) using Cohen's d; Test type: Other; Cohen's d = 0.36

3. Secondary Outcome: Test the Effect of tPBM on Impaired Decision Making
Description: Improvement in decision making will be evaluated by an increase in net gain at the Iowa Gambling Task (IGT) (higher score=better outcome, min score -3000, max score 7000), decrease in Barratt Impulsiveness Scale (BIS) score (min 30, max 120, lower score=better outcome), decrease in Behavior Rating Inventory of Executive Function - Adult Version (BRIEF-A) score (min 0, max 140, lower score=better outcome), and a decrease in I-7 Impulsiveness and Venturesomeness Questionnaire score (lower score=better outcome, Impulsiveness subscale: min 0, max 19, Venturesomeness subscale: min 0, max 15). All items are evaluated at Day 5 and Follow-up visit relative to Baseline. Baseline occurred approximately 1 week prior to Day 1. Treatment Days 2-5 were scheduled for the following week, ideally once daily, however the schedule allowed for flexibility, with Day 5 occurring no later than 10 days after Day 1. Follow-up occurred approximately 1 week after Day 5, or approximately 3 weeks after Baseline.
Time Frame: Baseline to Follow-Up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subjects
Number analyzed (Participants) | 4
units on a scale
  IGT Baseline | 3750 (805.19)
  IGT Day 1 | 4425 (448.14)
  IGT Day 5 | 4512.5 (586.48)
  IGT Follow-Up | 4637.5 (432.77)
  IGT Net Gain Baseline to Day 5 | 762.5 (228.67)
  BIS Baseline | 69.75 (8.77)
  BIS Day 5 | 70.5 (4.51)
  BIS Follow Up | 71.25 (8.01)
  BIS Change Baseline to Day 5 | 0.75 (5.38)
  BIS Change Baseline to Follow Up | 1.5 (8.22)
  BRIEF-A Baseline | 41.75 (27.18)
  BRIEF-A Day 5 | 58 (24.68)
  BRIEF-A Follow Up | 41.25 (24.53)
  BRIEF-A Change Baseline to Day 5 | 16.25 (25.86)
  BRIEF-A Change Baseline to Follow Up | -0.5 (4.12)
  I-7 Impulsiveness Baseline | 9.75 (5.31)
  I-7 Impulsiveness Day 5 | 9 (4.08)
  I-7 Impulsiveness Follow Up | 8.25 (3.59)
  I-7 Impulsiveness Change Baseline to Day 5 | -0.75 (2.99)
  I-7 Impulsiveness Change Baseline to Follow Up | -1.5 (2.38)
  I-7 Venturesomeness Baseline | 6.5 (3.51)
  I-7 Venturesomeness Day 5 | 6.25 (3.30)
  I-7 Venturesomeness Follow Up | 5.25 (3.77)
  I-7 Venturesomeness Change Baseline to Day 5 | -0.25 (1.26)
  I-7 Venturesomeness Change Baseline to Follow Up | -1.25 (0.96)
Statistical Analysis 1: Comparison: Subjects; The Wilcoxon signed-rank test was used to evaluate changes in the IGT at Baseline vs Day 5 due to the small sample size and distributional assumptions. Effect sizes were calculated using the rank biserial correlation coefficient (r) to estimate the magnitude of change; Test type: Other; p = 0.15, Wilcoxon signed rank test; rank biserial correlation coefficient = 0.767
Statistical Analysis 2: Comparison: Subjects; Test type: Other — The Friedman test was used to assess overall differences in IGT across Baseline, Day 1, and Day 5; p = 0.038, Friedman test
Statistical Analysis 3: Comparison: Subjects; Test type: Other — The Friedman test was used to assess overall differences in IGT across all timepoints (Baseline, Day 1, Day 5, Follow-Up); p = 0.043, Friedman test
Statistical Analysis 4: Comparison: Subjects; Test type: Other — The Wilcoxon signed-rank test was used to evaluate changes in the BIS across timepoints due to the small sample size and distributional assumptions. Effect sizes were calculated using the rank biserial correlation coefficient (r) to estimate the magnitude of change; p = 0.42, Wilcoxon signed rank test; BIS across timepoints; rank biserial correlation coefficient = 0.134
Statistical Analysis 5: Comparison: Subjects; Test type: Other — The Wilcoxon signed-rank test was used to evaluate changes in the BRIEF-A across timepoints due to the small sample size and distributional assumptions; p = 0.232, Wilcoxon signed rank test; BRIEF-A across timepoints
Statistical Analysis 6: Comparison: Subjects; Test type: Other — The Wilcoxon signed-rank test was used to evaluate changes in the i7 Impulsivity across timepoints due to the small sample size and distributional assumptions. Effect sizes were calculated using the rank biserial correlation coefficient (r) to estimate the magnitude of change; p = 0.06, Wilcoxon signed rank test; i7 Impulsivity; rank biserial correlation coefficient = 0.575
Statistical Analysis 7: Comparison: Subjects; Test type: Other — The Wilcoxon signed-rank test was used to evaluate changes in the i7 Venturesomeness across timepoints due to the small sample size and distributional assumptions. Effect sizes were calculated using the rank biserial correlation coefficient (r) to estimate the magnitude of change; p = 0.36, Wilcoxon signed rank test; rank biserial correlation coefficient = 0.275

4. Secondary Outcome: Test the Effect of Repeated t-PBM Sessions on Mood Symptoms (MOODS-SR) in Subjects With Bipolar Disorder (BD)
Description: Repeated t-PBM sessions on the rDLPFC will significantly decrease the total Mood Spectrum-Self Report (MOODS-SR) (min 0, max 154, lower score= better outcome) score at Day 5 and Follow-Up visit relative to Baseline. The scale was evaluated at Day 5 and Follow-up visit relative to Baseline. Baseline occurred approximately 1 week prior to Day 1. Treatment Days 2-5 were scheduled for the following week, ideally once daily, however the schedule allowed for flexibility, with Day 5 occurring no later than 10 days after Day 1. Follow-up occurred approximately 1 week after Day 5, or approximately 3 weeks after Baseline.
Time Frame: Baseline to Follow Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects
Number analyzed (Participants) | 4
score on a scale
  MOODS-SR Baseline | 18.5 (23.44)
  MOODS-SR Day 5 | 21.5 (26.41)
  MOODS-SR Follow Up | 13.5 (17.84)
  MOODS-SR Change Baseline to Day 5 | 3 (8.83)
  MOODS-SR Change Baseline to Follow Up | -5 (5.83)
Statistical Analysis 1: Comparison: Subjects; Test type: Other — Non-parametric tests were employed to evaluate changes across MOODS-SR Baseline to Day 5 due to the small sample size and distributional assumptions. The Wilcoxon signed-rank tests were applied for pairwise comparisons. Effect sizes were calculated using Cohen's d to estimate the magnitude of change; p = 0.6, Wilcoxon signed rank test; Cohen's d = 0.12
Statistical Analysis 2: Comparison: Subjects; Test type: Other — Non-parametric tests were employed to evaluate changes across MOODS-SR Baseline to Follow Up due to the small sample size and distributional assumptions. The Wilcoxon signed-rank tests were applied for pairwise comparisons. Effect sizes were calculated using Cohen's d to estimate the magnitude of change; p = 0.2, Wilcoxon signed rank test; Cohen's d = 0.24

ADVERSE EVENTS:
Time Frame: Adverse events were collected at all visits apart from screening (Baseline, Day 1-5, Follow Up). Adverse events were also collected during a clinician check-in between Day 5 and Follow Up, approximately 2-3 days after Day 5. Baseline occurred approximately 1 week prior to Day 1. Treatment Days 2-5 were scheduled for the following week (daily); the schedule allowed for flexibility, with Day 5 occurring no later than 10 days after Day 1. Follow-up occurred approximately 1 week after Day 5.
Description: The Adverse Events Form captures any adverse event (serious or otherwise) that the subject experiences while participating in the study. Events may occur during or outside of study procedures. Subjects or staff could report Adverse Events. The event, severity, resolution, relatedness to treatment, action taken, and expectedness were all documented along with the start and end date (course) of the Adverse Event.
Arm/Group | Subjects
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects (N=4)
Skin Warming (Skin and subcutaneous tissue disorders) | 3 (8) — Participant noted some slight skin warming during treatment.
Skin Reddening Under Diode (Skin and subcutaneous tissue disorders) | 3 (5) — Redness under diode sites post-treatment
Cold-like Virus/Common Cold (Infections and infestations) | 2 (2)
Pimple on Forehead at Diode Location (Skin and subcutaneous tissue disorders) | 1 (1) — Pimple on forehead at the F4 diode location. Identified at the end of the tx session. Ptp reported it is uncommon for her to get pimples on her forehead.
Visual Illusion (Psychiatric disorders) | 1 (1) — Brief visual illusion while biking to work. Participant reported she saw "a monster swiping out to get me" but then realized it was just a bike rack. Potential perception issue, visual perception or misperception.

LIMITATIONS AND CAVEATS:
The sample size is small, limiting statistical analyses and interpretation. The results highlight the need for group-level statistical analyses in a larger sample to validate. The inter-individual variability suggests that future studies should include additional longitudinal tracking and more examination of moderating factors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT05408637/Prot_SAP_000.pdf